CLINICAL TRIAL: NCT00123617
Title: The Impact of Cardiac Rehabilitation on Angina Frequency, Psychological Morbidity and Quality of Life in Women With Syndrome X
Brief Title: The Impact of Cardiac Rehabilitation Participation on Cardiac Syndrome X
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart and Lung Institute (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Prof. Peter Collins, Professor of Clinical Cardiology, National Heart and Lung Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-239
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Microvascular Angina
Keywords: Chest pain; Women; Syndrome X; Cardiac rehabilitation; Psychological morbidity; Cardiovascular risk factors
MeSH Terms: conditions — Microvascular Angina; Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase III cardiac rehabilitation (Experimental): Phase III group-based cardiac rehabilitation classes, weekly
  Interventions: Procedure: Phase III group-based cardiac rehabilitation
- Monitoring (No Intervention): Normal daily living, no extra visits to study centre

INTERVENTIONS:
Procedure: Phase III group-based cardiac rehabilitation — Phase III group-based cardiac rehabilitation
  Other Names: Cardiac rehab
  Arms: Phase III cardiac rehabilitation

SUMMARY:
The study is designed to test the hypothesis that participation in a standard phase III group based cardiac rehabilitation programme will improve psychological morbidity, quality of life and cardiovascular risk factors, along with chest pain severity and frequency in women with cardiac syndrome X.

DETAILED DESCRIPTION:
Very few clinicians treating patients with Syndrome X could dispute that despite an excellent prognosis, the debilitating symptomology and ineffective treatment regimes typical in this condition give patients a miserable quality of life. First identified by Kemp (1), the triad of angina pectoris, a positive exercise test for myocardial ischemia and angiographically smooth coronary arteries continues to perplex clinician seeking a useful treatment regime.

The possible pathophysiology of chest pain associated with Syndrome X is poorly understood in these patients. Suggested mechanisms include abnormal myocardial flow reserve due to coronary microvascular dysfunction ('microvascular angina') (2) or a generalised disorder of vascular function (3),(4) early signs of abnormal left ventricular function (5), which in some patients may deteriorate over time,(6) and abnormal visceral pain perception (7). Some patients exhibit insulin resistance (8). However, there have been few adequate systematic explorations of the psychological and social aspects of Syndrome X.

Several studies have found increased levels of anxiety in patients with normal or near normal coronary arteries in the presence of accompanying chest pain (9). Ruggeri et al (10) found higher level of neuroticism and anxiety in small group of patients with Syndrome X in comparison with patients with confirmed coronary artery disease. Panic disorders, sometimes associated with chest pain, are also often presented with depression, hypochondriasis or other somatoform disorders (11). Studies investigating various non-therapeutic treatment regimes have repeatedly shown that relaxation and stress reduction lead to fewer incidence of chest pain in Syndrome X patients (12). However, the same is also true for patients with CAD (13) along with many other conditions and disorders with related chronic pain (14).

Frequency and severity of chest pain has been shown to have a direct effect on quality of life in Syndrome X patients (15). Sand (16) found that over a 7-year follow-up, a higher percentage of Syndrome X patients had given up work, reduced their daily activities and reported worsening chest pain in comparison to patients with confirmed coronary disease. Persistent functional incapacity with concomitant high levels of chest pain in patients with normal or near normal coronary arteries was also found after an 11-year follow-up (9). Use of anti-anginals was higher, as was their self reported burden on the health service.

The Collins team recently performed the largest psychosocial investigation of postmenopausal women with Syndrome X ever undertaken (17). The Hearts and Minds Study, which involved 100 Syndrome X patients, 100 patients with CHD and 100 healthy volunteers found that Syndrome X patients suffered significantly higher levels of anxiety than CHD patients or healthy controls. A greater number of Syndrome X patients suffered clinical levels of anxiety and depression than CHD patients and healthy volunteers, along with suffering significantly higher levels of psychological suffering as measured by the Health Anxiety Questionnaire than healthy controls. We also found that Syndrome X patients with a small social network had higher levels of anxiety than their counterparts with a larger social support structure.

In order to address these findings, it is important to identify an intervention which not only reduces anxiety, but also promotes wellbeing, improves quality of life and augments the social support resource network available to Syndrome X patients. Cardiac Rehabilitation (CR) has consistently been shown to improve the psychological wellbeing in cardiac patients, as recent reviews have highlighted the beneficial effects of CR on symptoms of angina and dyspnoea, stress level and psychological functioning (18). CR has been shown to have a positive affect on reducing anxiety levels in cardiovascular patients (19), while high levels of depression, a frequent co-morbidity in MI patients, have been reduced by CR (20). Women in particular seem to gain most benefit from CR, as improvements in functional capacity, coronary risk and psychosocial wellbeing were equal or greater in women than men following rehabilitation (21). It has been suggested that CR may reduce anxiety in CHD patients by reducing uncertainty, providing patients with an optimistic yet realistic outlook of recovery, as well as providing psychological support and promoting coping (18). Few could argue that a similar outcome in Syndrome X patients would not be beneficial.

As well as promoting psychological wellbeing, CR also provides patients with a social support resource network. The adequacy of social support has been investigated in relation the prognosis of patients with CHD (22) when it was noted that inadequate tangible support was a significant predictor of both morbidity and mortality. Population based studies have consistently identified a link between social support and CHD morbidity and mortality in men, while disease severity and proliferation have been shown to be related to a lack of support in women (23). Epidemiological studies have also consistently found a link between depression, social isolation and predicted morbidity and mortality in CAD patients (24). It has been argued that CR provides the social context through which coronary prevention interventions are delivered (25) and that this extra social support may have an important part to play in the patients recovery from, and adaptation to, chronic illness (26).

The effect of exercise intervention on the frequency and severity of angina has been the object of investigation for many years. Some studies have reported a reduction in mean weekly episodes of angina of up to 91% using an acute exercise intervention in CHD patients (13) and while other studies have been unable to replicate such results, almost all highlight the beneficial effect of exercise on angina frequency. Nevertheless, very few studies have investigated the impact of exercise on Syndrome X, either from a psychosocial or physiological view-point. Erikkson et al (27) addressed the physical deconditioning apparent in many Syndrome X patients through the use of 8 weeks moderate intensity exercise. Time to pain improved dramatically, with no increase in maximum pain experienced, while peak exercise capacity, heart rate and systolic blood pressure also showed improvements. Exercise capacity and quality of life were also shown to increase following 8 weeks of physical training in separate group of Syndrome X patients (28).

Aerobic exercise has been repeatedly shown to have positive effects on psychological wellbeing, anxiety and depression (29). Patients suffering clinical levels of anxiety and depression have shown a reduction in the severity of their symptoms(30)while athletes and the very active became depressed when they were prevented from exercising(31). Studies involving exercise, anxiety and wellbeing the older population are limited, however subjective health and psychological wellbeing have been shown to be higher among older people who partake in regular exercise (32). Anxiety reduction and increased wellbeing has also been shown in elderly men following an 8-week weekly exercise intervention (33).

Therefore, we would like to explore the beneficial effects of cardiac rehabilitation in Syndrome X patients. Exercise is not currently recognised as a treatment regime for Syndrome X, either as a stand- alone intervention or in conjunction with any other therapy. Patients are currently given little advice or guidance relating to physical activity due to the lack of research and information regarding the potential benefit of exercise available to practitioners. Our previous investigations of Syndrome X have demonstrated a need for an intervention which would not only reduce the patients reported levels of anxiety, but also increase their perceived social support, psychological wellbeing and quality of life. CR has been shown to improve quality of life, reduce anxiety and decrease frequency of angina episodes in CHD patients through the use of exercise intervention and tangible social support. Therefore, we would like to investigate the following research questions:

Does cardiac rehabilitation:

1. Reduce the frequency and severity of angina attacks in Syndrome X?
2. Reduce anxiety, depression and health related worry found in Syndrome X?
3. Improve the quality of life of Syndrome X patients?

Reference List

1. Kemp HG, Jr., Vokonas PS, Cohn PF, Gorlin R. The anginal syndrome associated with normal coronary arteriograms. Report of a six year experience. Am J Med 1973; 54(6):735-742.
2. Cannon RO, III, Epstein SE. "Microvascular angina" as a cause of chest pain with angiographically normal coronary arteries. Am J Cardiol 1988; 61(15):1338-1343.
3. Raymond C. Chest pain not always what it seems; panic disorder may be cause in some. JAMA 1989; 261(8):1101-1102.
4. Sax FL, Cannon RO, III, Hanson C, Epstein SE. Impaired forearm vasodilator reserve in patients with microvascular angina. Evidence of a generalized disorder of vascular function? N Engl J Med 1987; 317(22):1366-1370.
5. Cannon RO, III, Bonow RO, Bacharach SL, Green MV, Rosing DR, Leon MB et al. Left ventricular dysfunction in patients with angina pectoris, normal epicardial coronary arteries, and abnormal vasodilator reserve. Circulation 1985; 71(2):218-226.
6. Opherk D, Schuler G, Wetterauer K, Manthey J, Schwarz F, Kubler W. Four-year follow-up study in patients with angina pectoris and normal coronary arteriograms ("syndrome X"). Circulation 1989; 80(6):1610-1616.
7. Shapiro LM, Crake T, Poole-Wilson PA. Is altered cardiac sensation responsible for chest pain in patients with normal coronary arteries? Clinical observation during cardiac catheterisation. Br Med J (Clin Res Ed) 1988; 296(6616):170-171.
8. Dean JD, Jones CJ, Hutchison SJ, Peters JR, Henderson AH. Hyperinsulinaemia and microvascular angina ("syndrome X"). Lancet 1991; 337(8739):456-457.
9. Potts SG, Bass CM. Psychological morbidity in patients with chest pain and normal or near- normal coronary arteries: a long-term follow-up study . Psychol Med 1995; 25(2):339-347.
10. Ruggeri A, Taruschio G, Loricchio ML, Samory G, Borghi A, Bugiardini R. [The correlation between the clinical characteristics and psychological status in syndrome X patients]. Cardiologia 1996; 41(6):551-557.
11. Mayou R. Chest pain, palpitations and panic. J Psychosom Res 1998; 44(1):53-70.
12. Cunningham C, Brown S, Kaski JC. Effects of transcendental meditation on symptoms and electrocardiographic changes in patients with cardiac syndrome X. Am J Cardiol 2000; 85(5):653-5, A10.
13. Ornish D, Scherwitz LW, Doody RS, Kesten D, McLanahan SM, Brown SE et al. Effects of stress management training and dietary changes in treating ischemic heart disease. JAMA 1983; 249(1):54-59.
14. Luebbert K, Dahme B, Hasenbring M. The effectiveness of relaxation training in reducing treatment-related symptoms and improving emotional adjustment in acute non-surgical cancer treatment: a meta-analytical review. Psychooncology 2001; 10(6):490-502.
15. Atienza F, Velasco JA, Brown S, Ridocci F, Kaski JC. Assessment of quality of life in patients with chest pain and normal coronary arteriogram (syndrome X) using a specific questionnaire. Clin Cardiol 1999; 22(4):283-290.
16. Sand NP, Juelsgaard P. [Syndrome X. Somatic and social prognosis of patients with angina pectoris and normal coronary arteriography]. Ugeskr Laeger 1994; 156(8):1131-1136.
17. Asbury EA, Creed F, Collins P. Distinct psychosocial differences between women with coronary heart disease and cardiac syndrome X. Eur Heart J 2004; 25 (19):1695-1701.
18. Grace SL, Abbey SE, Shnek ZM, Irvine J, Franche RL, Stewart DE. Cardiac rehabilitation I. review of psychosocial factors. Gen Hosp Psychiatry 2002; 24(3):121-126.
19. Yoshida T, Kohzuki M, Yoshida K, Hiwatari M, Kamimoto M, Yamamoto C et al. Physical and psychological improvements after phase II cardiac rehabilitation in patients with myocardial infarction. Nurs Health Sci 1999; 1(3):163-170.
20. Johnston M, Foulkes J, Johnston DW, Pollard B, Gudmundsdottir H. Impact on patients and partners of inpatient and extended cardiac counseling and rehabilitation: a controlled trial. Psychosom Med 1999; 61(2):225-233.
21. O'Callaghan WG, Teo KK, O'Riordan J, Webb H, Dolphin T, Horgan JH. Comparative response of male and female patients with coronary artery disease to exercise rehabilitation. Eur Heart J 1984; 5(8):649-651.
22. Woloshin S, Schwartz LM, Tosteson AN, Chang CH, Wright B, Plohman J et al. Perceived adequacy of tangible social support and health outcomes in patients with coronary artery disease. J Gen Intern Med 1997; 12(10):613-618.
23. Horsten M, Mittleman MA, Wamala SP, Schenck-Gustafsson K, Orth-Gomer K. Depressive symptoms and lack of social integration in relation to prognosis of CHD in middle-aged women. The Stockholm Female Coronary Risk Study. Eur Heart J 2000; 21(13):1072-1080.
24. Wenger NK. Social support and coronary heart disease in women: the challenge to learn more. Eur Heart J 1998; 19(11):1603-1605.
25. Lindsay GM, Smith LN, Hanlon P, Wheatley DJ. The influence of general health status and social support on symptomatic outcome following coronary artery bypass grafting. Heart 2001; 85(1):80-86.
26. Anderson D, Deshaies G, Jobin J. Social support, social networks and coronary artery disease rehabilitation: a review. Can J Cardiol 1996; 12(8):739-744.
27. Eriksson BE, Tyni-Lenne R, Svedenhag J, Hallin R, Jensen-Urstad K, Jensen-Urstad M et al. Physical training in Syndrome X: physical training counteracts deconditioning and pain in Syndrome X. J Am Coll Cardiol 2000; 36(5):1619-1625.
28. Tyni-Lenne R, Stryjan S, Eriksson B, Berglund M, Sylven C. Beneficial therapeutic effects of physical training and relaxation therapy in women with coronary syndrome X. Physiother Res Int 2002; 7(1):35-43.
29. Salmon P. Effects of physical exercise on anxiety, depression, and sensitivity to stress: a unifying theory. Clin Psychol Rev 2001; 21(1):33-61.
30. Craft LL, Landers D.M. The effect of exercise on clinical depression and depression resulting from mental illness: A meta analysis. Journal of Sport and Exercise Psychology 20, 339-357. 1998.
31. Aidman EV, Woollard S. The influence of self-reported exercise addiction on acute emotional and physiological responses to brief exercise deprivation. Psychology of Sport and Exercise. 2002.
32. Ransford HE, Palisi BJ. Aerobic exercise, subjective health and psychological well-being within age and gender subgroups. Soc Sci Med 1996; 42(11):1555-1559.
33. Perrig-Chiello P, Perrig WJ, Ehrsam R, Staehelin HB, Krings F. The effects of resistance training on well-being and memory in elderly volunteers. Age Ageing 1998; 27(4):469-475.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Aged 30 to 80 years
* Postmenopausal > 1 year since last menstrual period
* Angiographically normal coronary arteries
* Positive treadmill exercise test for myocardial ischemia
* Reported angina pectoris > 2 episodes per week
* Diagnosis > 6 months
* Willing to give written informed consent

Exclusion Criteria:

* History of psychiatric illness
* History of any other chronic illness
* Participation in another research study within the previous 60 days
* Suffer any physical condition for which exercise is a contra-indication.
* Unwilling to give written informed consent

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2003-01; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Anxiety | Measured at baseline then every 8 weeks for 16 weeks
Depression | Measured at baseline then every 8 weeks for 16 weeks
Health anxiety | Measured at baseline then every 8 weeks for 16 weeks
Cardiac anxiety | Measured at baseline then every 8 weeks for 16 weeks
Quality of life | Measured at baseline then every 8 weeks for 16 weeks
Symptom severity | Measured at baseline then continuously for 16 weeks
Symptom frequency | Measured at baseline then continuously for 16 weeks

SECONDARY OUTCOMES:
Cardiovascular risk factors | Measured at baseline, 8 weeks and 16 weeks.
Physical ability | Baseline and at 8 weeks
Time to pain | Baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Collins, MD FRCP, Principal Investigator — National Heart and Lung Institute, Imperial College London
Locations (1):
- National Heart and Lung Institute, Imperial College London, London, United Kingdom

REFERENCES:
- [Background] Kemp HG Jr, Vokonas PS, Cohn PF, Gorlin R. The anginal syndrome associated with normal coronary arteriograms. Report of a six year experience. Am J Med. 1973 Jun;54(6):735-42. doi: 10.1016/0002-9343(73)90060-0. No abstract available. PMID 4196179
- [Background] Cannon RO 3rd, Epstein SE. "Microvascular angina" as a cause of chest pain with angiographically normal coronary arteries. Am J Cardiol. 1988 Jun 1;61(15):1338-43. doi: 10.1016/0002-9149(88)91180-0. No abstract available. PMID 3287885
- [Background] Raymond C. Chest pain not always what it seems; panic disorder may be cause in some. JAMA. 1989 Feb 24;261(8):1101-2. No abstract available. PMID 2915426
- [Background] Sax FL, Cannon RO 3rd, Hanson C, Epstein SE. Impaired forearm vasodilator reserve in patients with microvascular angina. Evidence of a generalized disorder of vascular function? N Engl J Med. 1987 Nov 26;317(22):1366-70. doi: 10.1056/NEJM198711263172202. PMID 3683470
- [Background] Cannon RO 3rd, Bonow RO, Bacharach SL, Green MV, Rosing DR, Leon MB, Watson RM, Epstein SE. Left ventricular dysfunction in patients with angina pectoris, normal epicardial coronary arteries, and abnormal vasodilator reserve. Circulation. 1985 Feb;71(2):218-26. doi: 10.1161/01.cir.71.2.218. PMID 3965167
- [Background] Opherk D, Schuler G, Wetterauer K, Manthey J, Schwarz F, Kubler W. Four-year follow-up study in patients with angina pectoris and normal coronary arteriograms ("syndrome X"). Circulation. 1989 Dec;80(6):1610-6. doi: 10.1161/01.cir.80.6.1610. PMID 2598425
- [Background] Shapiro LM, Crake T, Poole-Wilson PA. Is altered cardiac sensation responsible for chest pain in patients with normal coronary arteries? Clinical observation during cardiac catheterisation. Br Med J (Clin Res Ed). 1988 Jan 16;296(6616):170-1. doi: 10.1136/bmj.296.6616.170-a. No abstract available. PMID 3122985
- [Background] Dean JD, Jones CJ, Hutchison SJ, Peters JR, Henderson AH. Hyperinsulinaemia and microvascular angina ("syndrome X"). Lancet. 1991 Feb 23;337(8739):456-7. PMID 1671472
- [Background] Potts SG, Bass CM. Psychological morbidity in patients with chest pain and normal or near-normal coronary arteries: a long-term follow-up study. Psychol Med. 1995 Mar;25(2):339-47. doi: 10.1017/s0033291700036242. PMID 7675922
- [Background] Ruggeri A, Taruschio G, Loricchio ML, Samory G, Borghi A, Bugiardini R. [The correlation between the clinical characteristics and psychological status in syndrome X patients]. Cardiologia. 1996 Jun;41(6):551-7. Italian. PMID 8766418
- [Background] Mayou R. Chest pain, palpitations and panic. J Psychosom Res. 1998 Jan;44(1):53-70. doi: 10.1016/s0022-3999(97)00209-2. PMID 9483464
- [Background] Cunningham C, Brown S, Kaski JC. Effects of transcendental meditation on symptoms and electrocardiographic changes in patients with cardiac syndrome X. Am J Cardiol. 2000 Mar 1;85(5):653-5, A10. doi: 10.1016/s0002-9149(99)00828-0. PMID 11078284
- [Background] Ornish D, Scherwitz LW, Doody RS, Kesten D, McLanahan SM, Brown SE, DePuey E, Sonnemaker R, Haynes C, Lester J, McAllister GK, Hall RJ, Burdine JA, Gotto AM Jr. Effects of stress management training and dietary changes in treating ischemic heart disease. JAMA. 1983 Jan 7;249(1):54-9. PMID 6336794
- [Background] Luebbert K, Dahme B, Hasenbring M. The effectiveness of relaxation training in reducing treatment-related symptoms and improving emotional adjustment in acute non-surgical cancer treatment: a meta-analytical review. Psychooncology. 2001 Nov-Dec;10(6):490-502. doi: 10.1002/pon.537. PMID 11747061
- [Background] Atienza F, Velasco JA, Brown S, Ridocci F, Kaski JC. Assessment of quality of life in patients with chest pain and normal coronary arteriogram (syndrome X) using a specific questionnaire. Clin Cardiol. 1999 Apr;22(4):283-90. doi: 10.1002/clc.4960220406. PMID 10198738
- [Background] Sand NP, Juelsgaard P. [Syndrome X. Somatic and social prognosis of patients with angina pectoris and normal coronary arteriography]. Ugeskr Laeger. 1994 Feb 21;156(8):1131-2, 1135-6. Danish. PMID 8116091
- [Background] Grace SL, Abbey SE, Shnek ZM, Irvine J, Franche RL, Stewart DE. Cardiac rehabilitation I: review of psychosocial factors. Gen Hosp Psychiatry. 2002 May-Jun;24(3):121-6. doi: 10.1016/s0163-8343(02)00178-0. PMID 12062135
- [Background] Yoshida T, Kohzuki M, Yoshida K, Hiwatari M, Kamimoto M, Yamamoto C, Meguro S, Endo N, Kato A, Kanazawa M, Sato T. Physical and psychological improvements after phase II cardiac rehabilitation in patients with myocardial infarction. Nurs Health Sci. 1999 Sep;1(3):163-70. doi: 10.1046/j.1442-2018.1999.00021.x. PMID 10894639
- [Background] Johnston M, Foulkes J, Johnston DW, Pollard B, Gudmundsdottir H. Impact on patients and partners of inpatient and extended cardiac counseling and rehabilitation: a controlled trial. Psychosom Med. 1999 Mar-Apr;61(2):225-33. doi: 10.1097/00006842-199903000-00015. PMID 10204976
- [Background] O'Callaghan WG, Teo KK, O'Riordan J, Webb H, Dolphin T, Horgan JH. Comparative response of male and female patients with coronary artery disease to exercise rehabilitation. Eur Heart J. 1984 Aug;5(8):649-51. doi: 10.1093/oxfordjournals.eurheartj.a061721. PMID 6479192
- [Background] Woloshin S, Schwartz LM, Tosteson AN, Chang CH, Wright B, Plohman J, Fisher ES. Perceived adequacy of tangible social support and health outcomes in patients with coronary artery disease. J Gen Intern Med. 1997 Oct;12(10):613-8. doi: 10.1046/j.1525-1497.1997.07121.x. PMID 9346457
- [Background] Horsten M, Mittleman MA, Wamala SP, Schenck-Gustafsson K, Orth-Gomer K. Depressive symptoms and lack of social integration in relation to prognosis of CHD in middle-aged women. The Stockholm Female Coronary Risk Study. Eur Heart J. 2000 Jul;21(13):1072-80. doi: 10.1053/euhj.1999.2012. PMID 10843825
- [Background] Wenger NK. Social support and coronary heart disease in women: the challenge to learn more. Eur Heart J. 1998 Nov;19(11):1603-5. No abstract available. PMID 9857910
- [Background] Lindsay GM, Smith LN, Hanlon P, Wheatley DJ. The influence of general health status and social support on symptomatic outcome following coronary artery bypass grafting. Heart. 2001 Jan;85(1):80-6. doi: 10.1136/heart.85.1.80. PMID 11119470
- [Background] Anderson D, Posner N. Relationship between psychosocial factors and health behaviours for women experiencing menopause. Int J Nurs Pract. 2002 Oct;8(5):265-73. doi: 10.1046/j.1440-172x.2002.00376.x. PMID 12225353
- [Background] Eriksson BE, Tyni-Lenne R, Svedenhag J, Hallin R, Jensen-Urstad K, Jensen-Urstad M, Bergman K, Selven C. Physical training in Syndrome X: physical training counteracts deconditioning and pain in Syndrome X. J Am Coll Cardiol. 2000 Nov 1;36(5):1619-25. doi: 10.1016/s0735-1097(00)00931-1. PMID 11079667
- [Background] Tyni-Lenne R, Stryjan S, Eriksson B, Berglund M, Sylven C. Beneficial therapeutic effects of physical training and relaxation therapy in women with coronary syndrome X. Physiother Res Int. 2002;7(1):35-43. doi: 10.1002/pri.239. PMID 11992983
- [Background] Salmon P. Effects of physical exercise on anxiety, depression, and sensitivity to stress: a unifying theory. Clin Psychol Rev. 2001 Feb;21(1):33-61. doi: 10.1016/s0272-7358(99)00032-x. PMID 11148895
- [Background] Ransford HE, Palisi BJ. Aerobic exercise, subjective health and psychological well-being within age and gender subgroups. Soc Sci Med. 1996 Jun;42(11):1555-9. doi: 10.1016/0277-9536(95)00252-9. PMID 8771638
- [Background] Perrig-Chiello P, Perrig WJ, Ehrsam R, Staehelin HB, Krings F. The effects of resistance training on well-being and memory in elderly volunteers. Age Ageing. 1998 Jul;27(4):469-75. doi: 10.1093/ageing/27.4.469. PMID 9884004
- [Result] Asbury EA, Slattery C, Grant A, Evans L, Barbir M, Collins P. Cardiac rehabilitation for the treatment of women with chest pain and normal coronary arteries. Menopause. 2008 May-Jun;15(3):454-60. doi: 10.1097/gme.0b013e31815982eb. PMID 18188136